CLINICAL TRIAL: NCT00831623
Title: Phase I-II Trial of Hypofractionated Conformal Proton Beam Radiation Therapy for Favorable-risk Prostate Cancer
Brief Title: Study of Hypofractionated Proton Beam Radiation Therapy for Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Jerry D. Slater, MD, Professor and Chair Department of Radiation Medicine, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 58116
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Results first posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer
Keywords: hypofractionation; proton beam radiation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Proton Therapy; Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Proton radiation therapy (Experimental): Single arm
  Interventions: Radiation: Proton Radiation; Radiation: Proton

INTERVENTIONS:
Radiation: Proton Radiation — 3 Cobalt Gray Equivalent (CGE) /Day to isocenter, one treatment per day, 5 days per week for 20 treatments (=60 CGE to isocenter/20 fractions)
Radiation: Proton — As above
  Other Names: Proton Radiation treatment

SUMMARY:
The purpose of this study is to determine hypofractionated conformal proton beam radiation therapy of prostate cancer can achieve similar treatment benefits as our current institutional standard with conventional fractionation.

DETAILED DESCRIPTION:
Radiation therapy has a long and established role in the curative treatment of organ-confined prostate cancer. However, the optimal radiation dose and treatment schedule remain unknown. The use of hypofractionation has a long and generally successful history in conformal proton beam therapy. Several reports detailing the efficacy and safety of hypofractionated conformal radiation therapy (with x-rays) of prostate cancer can be found in the literature. Hypofractionated conformal proton beam radiation therapy has become our institutional routine for the treatment of numerous solid tumors. The purpose of this study is to determine if a shortened overall treatment schedule will result in equivalent tumor control rates and no increased side effects as compared to our current institutional standard treatment of an equivalent dose given over a longer period of time.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma within 180 days of registration
* History & Physical Exam, including digital rectal exam (DRE), within 8 wks prior to registration
* Histologic evaluation of prostate biopsies at LLUMC, with Gleason score assignment
* Clinical stage, Tumor Stage (T1-T2C)
* Prostatic Specific Antigen (PSA) less than 10 ng.ml within 180 days prior to registration

Exclusion Criteria:

* Prior or concurrent invasive malignancy
* Evidence of distant metastasis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Treatment for prostate cancer in males
Enrollment: 167 (Actual)
Dates: Start 2009-02-17 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry D Slater, MD, Principal Investigator — Loma Linda University Medical Center Dept. of Radiation Medicine
Locations (1):
- Loma Linda University Medical Center / James M. Slater Proton Treatment Center, Loma Linda, California, United States

REFERENCES:
- [Background] Zietman AL, DeSilvio ML, Slater JD, Rossi CJ Jr, Miller DW, Adams JA, Shipley WU. Comparison of conventional-dose vs high-dose conformal radiation therapy in clinically localized adenocarcinoma of the prostate: a randomized controlled trial. JAMA. 2005 Sep 14;294(10):1233-9. doi: 10.1001/jama.294.10.1233. PMID 16160131
- [Background] Rossi CJ Jr, Slater JD, Yonemoto LT, Jabola BR, Bush DA, Levy RP, Grove R, Slater JM. Influence of patient age on biochemical freedom from disease in patients undergoing conformal proton radiotherapy of organ-confined prostate cancer. Urology. 2004 Oct;64(4):729-32. doi: 10.1016/j.urology.2004.04.043. PMID 15491710
- [Background] Slater JD, Rossi CJ Jr, Yonemoto LT, Bush DA, Jabola BR, Levy RP, Grove RI, Preston W, Slater JM. Proton therapy for prostate cancer: the initial Loma Linda University experience. Int J Radiat Oncol Biol Phys. 2004 Jun 1;59(2):348-52. doi: 10.1016/j.ijrobp.2003.10.011. PMID 15145147
- [Background] Slater JM, Bush DA, Grove R, Slater JD. The prognostic value of percentage of positive biopsy cores, percentage of cancer volume, and maximum involvement of biopsy cores in prostate cancer patients receiving proton and photon beam therapy. Technol Cancer Res Treat. 2014 Jun;13(3):227-31. doi: 10.7785/tcrtexpress.2013.600271. Epub 2013 Sep 20. PMID 24066950
- [Background] Coen JJ, Bae K, Zietman AL, Patel B, Shipley WU, Slater JD, Rossi CJ. Acute and late toxicity after dose escalation to 82 GyE using conformal proton radiation for localized prostate cancer: initial report of American College of Radiology Phase II study 03-12. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):1005-9. doi: 10.1016/j.ijrobp.2010.06.047. Epub 2010 Oct 6. PMID 20932675
- [Background] Talcott JA, Rossi C, Shipley WU, Clark JA, Slater JD, Niemierko A, Zietman AL. Patient-reported long-term outcomes after conventional and high-dose combined proton and photon radiation for early prostate cancer. JAMA. 2010 Mar 17;303(11):1046-53. doi: 10.1001/jama.2010.287. PMID 20233822
- [Background] Zietman AL, Bae K, Slater JD, Shipley WU, Efstathiou JA, Coen JJ, Bush DA, Lunt M, Spiegel DY, Skowronski R, Jabola BR, Rossi CJ. Randomized trial comparing conventional-dose with high-dose conformal radiation therapy in early-stage adenocarcinoma of the prostate: long-term results from proton radiation oncology group/american college of radiology 95-09. J Clin Oncol. 2010 Mar 1;28(7):1106-11. doi: 10.1200/JCO.2009.25.8475. Epub 2010 Feb 1. PMID 20124169
- [Background] Slater JD. Clinical applications of proton radiation treatment at Loma Linda University: review of a fifteen-year experience. Technol Cancer Res Treat. 2006 Apr;5(2):81-9. doi: 10.1177/153303460600500202. PMID 16551128
- [Background] Ronson BB, Yonemoto LT, Rossi CJ, Slater JM, Slater JD. Patient tolerance of rectal balloons in conformal radiation treatment of prostate cancer. Int J Radiat Oncol Biol Phys. 2006 Apr 1;64(5):1367-70. doi: 10.1016/j.ijrobp.2005.11.001. Epub 2006 Feb 20. PMID 16488552
- [Background] Slater JD, Rossi CJ Jr, Yonemoto LT, Reyes-Molyneux NJ, Bush DA, Antoine JE, Miller DW, Teichman SL, Slater JM. Conformal proton therapy for early-stage prostate cancer. Urology. 1999 May;53(5):978-84. doi: 10.1016/s0090-4295(99)00014-x. PMID 10223493
- [Background] Slater JD, Yonemoto LT, Rossi CJ Jr, Reyes-Molyneux NJ, Bush DA, Antoine JE, Loredo LN, Schulte RW, Teichman SL, Slater JM. Conformal proton therapy for prostate carcinoma. Int J Radiat Oncol Biol Phys. 1998 Sep 1;42(2):299-304. doi: 10.1016/s0360-3016(98)00225-9. PMID 9788407
- [Background] Slater JD. Twenty years of proton radiation therapy at Loma Linda University Medical Center. In U. Linz, editor. Ion beam therapy: fundamentals, technology, clinical applications. Berlin: Springer, 2012:581-595.
- [Result] Slater JM, Slater JD, Kang JI, Namihas IC, Jabola BR, Brown K, Grove R, Watt C, Bush DA. Hypofractionated Proton Therapy in Early Prostate Cancer: Results of a Phase I/II Trial at Loma Linda University. Int J Part Ther. 2019 Summer;6(1):1-9. doi: 10.14338/IJPT-19-00057. Epub 2019 Aug 6. PMID 31773043

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Proton Radiation Therapy
Started | 167
Treated Per Protocol | 158
At Least 2 Years Since Completing Treatment | 146
Completed (At least two years since completing treatment) | 145
Not Completed | 22
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 1
Not completed — Not 2 years post-treatment | 12

BASELINE CHARACTERISTICS:
Population: 8 refused treatment, 158 treated per protocol, 146 at least 2 years since completing treatment, 1 with no follow up data
Groups:
- Study of Hypofractionated Proton Beam Radiation Therapy for Prostate Cancer: Patients with localized prostate cancer with the following characteristics:
  * Histologically confirmed adenocarcinoma within 180 days of registration
  * History & Physical Exam, including digital rectal exam (DRE), within 8 wks prior to registration
  * Histologic evaluation of prostate biopsies at LLUMC, with Gleason score assignment
  * Clinical stage, Tumor Stage (T1-T2C)
  * Prostatic Specific Antigen (PSA) less than 10 ng.ml within 180 days prior to registration
Arm/Group | Study of Hypofractionated Proton Beam Radiation Therapy for Prostate Cancer
Number analyzed (Participants) | 146
Age, Categorical [Count of Participants; unit: Participants] — Population: 8 refused treatment, 158 treated per protocol, 146 at least 2 years since completing treatment, 1 with no follow up data
  Participants
    <=18 years | 0
    Between 18 and 65 years | 70
    >=65 years | 76
Age, Continuous [Median (Full Range); unit: Years] — Population: 8 refused treatment, 158 treated per protocol, 146 at least 2 years since completing treatment, 1 with no follow up data
  Years | 65 [33 to 80]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 146
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 146
PSA [Median (Full Range); unit: ng/mL] | 4.98 [0.3 to 10.2]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Late Treatment-Related Toxicity Greater Than or Equal to Grade 3, CTCAE Version 4.0
Description: To determine if late CTCAE version 4.0 Grade 3 treatment-related morbidity, which is no worse than that engendered by our current institutional standard with conventional fractionation, can be maintained in a hypofractionated schedule.
Time Frame: Every 6 months after completing treatment through the duration of the trial with a minimum of 2 years follow-up and an average of 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Radiation Therapy
Number analyzed (Participants) | 146
Participants | 1

2. Secondary Outcome: Number of Participants With Acute and Late Gastrointestinal or Genitourinary Grade 2 Morbidity, CTCAE Version 4.0
Description: To determine if late CTCAE version 4.0 Grade 2 treatment-related morbidity, which is no worse than that engendered by our current institutional standard with conventional fractionation, can be maintained in a hypofractionated schedule.
Time Frame: Every 6 months after completing treatment through the duration of the trial, with a minimum of 2 years follow-up and an average of 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Radiation Therapy
Number analyzed (Participants) | 146
Participants | 21

ADVERSE EVENTS:
Time Frame: Patients toxicity was assessed at 6 month intervals following completion of treatment through the duration of the trial for a minimum of 2 years, with an average of 5 years.
Description: Acute toxicity was defined as toxicity during treatment and within the three-month post-treatment time point. Late toxicity was defined as toxicity occurring greater than three months post-treatment. Follow-up visits were conducted every three months for the first two years after treatment, every six months for the next three years, and annually thereafter. During follow-up visits history and physical exam were performed, PSA was measured, and toxicity was evaluated.
Arm/Group | Proton Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 0/146
Serious Adverse Events (participants affected / at risk) | 1/146
Other Adverse Events (participants affected / at risk) | 20/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Radiation Therapy (N=146)
Hematuria (Renal and urinary disorders) | 1 (1) — Gross hematuria in a patient with a long history of nephrolithiasis, and had nephrolithiasis found on cystoscopy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Radiation Therapy (N=146)
Grade 2 Gastrointestinal toxicity (Gastrointestinal disorders) | 7 (7) — incidence of grade 2 gastrointestinal toxicity was 4%
Grade 2 Genitourinary toxicity (Renal and urinary disorders) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-11-21): https://cdn.clinicaltrials.gov/large-docs/23/NCT00831623/Prot_SAP_000.pdf
  • Informed Consent Form (2015-05-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT00831623/ICF_001.pdf